CLINICAL TRIAL: NCT00582504
Title: A Phase 2 Open-Label, Safety and Immunogenicity Study of a Single Dose of Venezuelan Equine Encephalomyelitis Vaccine, Live, Attenuated, Dried, TC-83, NDBR-102, as Primary Immunization in Healthy Adults At Risk for Exposure to Virulent Venezuelan Equine Encephalomyelitis Virus
Brief Title: Safety and Immunogenicity Study of the Venezuelan Equine Encephalomyelitis Vaccine
Acronym: VEE TC-83
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-14317; FY06-26 (Other: IRB)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Venezuelan Equine Encephalomyelitis
Keywords: Encephalitis,VEE
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccination (Experimental): VEE TC-83
  Interventions: Biological: VEE TC-83

INTERVENTIONS:
Biological: VEE TC-83 — Subjects will receive a single 0.5 mL dose by subcutaneous route in the upper outer aspect of arm

SUMMARY:
This study is designed to determine safety of and immune response to Venezuelan Equine Encephalomyelitis Vaccine, Live, Attenuated, Dried TC-83, NDBR-102 (TC-83).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* VEE PRNT80 < 1:10 before immunization.
* (females) Negative serum pregnancy test on same day before vaccination. Not planning pregnancy for 3 months.
* Actively enrolled in the SIP
* At risk for exposure to virulent VEE virus (with up-to-date risk assessment).
* Up-to-date (within 1 year) physical examination/tests.
* Sign and date the approved informed consent.
* Willing to return for all follow-up visits.
* Agree to report adverse event (AE) up to 28 days after vaccination.

Exclusion Criteria:

* Over age of 65 years.
* Clinically significant abnormal lab results including evidence of Hepatitis C, Hepatitis B carrier state, or elevated liver function tests.
* History of immunodeficiency or current treatment with immunosuppressive medication.
* (females) Currently breastfeeding.
* Confirmed human immunodeficiency virus (HIV) titer.
* Family history (first degree relative, but not elderly parent with late onset) diabetes, personal history gestational diabetes, or confirmed elevated fasting serum glucose (> 125 mg/dL).
* Serious allergic reaction to guinea pigs/guinea pig products.
* Any known allergies to components of the vaccine.
* A medical condition that in the judgment of the Principal Investigator (PI) would impact subject safety (i.e-vaccination and or exposure to another alphavirus).
* Administration of any vaccine within 28 days of TC-83.
* Any unresolved AEs resulting from a previous immunization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a 80% plaque-reduction neutralization titer (PRNT80) | 21-35 days, 42-56 days, 12-15 months
Number of adverse events. | 7 years

SECONDARY OUTCOMES:
Number of confirmed cases of VEE disease among vaccinated subjects who achieved a PRNT 80 ≥ 1:20. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Reisler, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States